CLINICAL TRIAL: NCT02293668
Title: Outcome of Three Controlled Ovarian Hyperstimulation Protocols in Poor Responding Infertility Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ercan Bastu, Associate Professor of Obstetrics and Gynecology, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: poor responders
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Combined 450 (Active Comparator): Recombinant FSH 225IU/day and human menopausal gonadotropin (hMG) 225IU/day will be initiated on the second or third day of spontaneous menstruation and continued until the day of ovulation triggering. Ovulation triggering will be performed with the administration of 10000IU of human chorionic gonadotropin (hCG) as soon as two-three follicles of 17 mm diameter will be observed by transvaginal ultrasound.
  Interventions: Drug: FSH 225IU and hMG 225IU
- Combined 300 (Active Comparator): Recombinant FSH 150IU/day and human menopausal gonadotropin (hMG) 150IU/day will be initiated on the second or third day of spontaneous menstruation and continued until the day of ovulation triggering. Ovulation triggering will be performed with the administration of 10000IU of human chorionic gonadotropin (hCG) as soon as two-three follicles of 17 mm diameter will be observed by transvaginal ultrasound.
  Interventions: Drug: FSH 150IU and hMG 150IU
- Letrozole and hMG (Active Comparator): Letrozole (Femara; Novartis, East Hanover, NJ) at a dose of 5 mg/day and human menopausal gonadotropin (hMG) 150IU/day will be initiated on the second or third day of spontaneous menstruation and continued until the day of ovulation triggering. Ovulation triggering will be performed with the administration of 10000 IU of human chorionic gonadotropin (hCG) as soon as two-three follicles of 17 mm diameter will be observed by transvaginal ultrasound.
  Interventions: Drug: Letrozole 5mg and hMG 150IU

INTERVENTIONS:
Drug: FSH 225IU and hMG 225IU
  Arms: Combined 450
Drug: FSH 150IU and hMG 150IU
  Arms: Combined 300
Drug: Letrozole 5mg and hMG 150IU
  Arms: Letrozole and hMG

SUMMARY:
There are different controlled ovarian hyperstimulation protocols utilized in infertility patients. In this study, our aim is to specifically compare three protocols in poor responding infertility patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible if they are poor ovarian responders according to the Bologna criteria (Ferraretti et al., 2011).
* Two out of three of the following criteria are essential in order to classify a patient as poor ovarian responder:

  * advanced maternal age (≥40 years) or any other risk factor for poor ovarian response;
  * a poor ovarian response (≤3 oocytes with a conventional stimulation protocol); or
  * an abnormal ovarian reserve test (antral follicle count, <7 follicles or anti-Mullerian hormone, <1.1 ng/ml).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 8 weeks

SECONDARY OUTCOMES:
Number of oocytes retrieved | 4 weeks
Number of transferable embryos | 4 weeks
Biochemical pregnancy rate | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University School of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041